CLINICAL TRIAL: NCT01394341
Title: Safety and Effect of Liraglutide in Patients With Type 2 Diabetes and Severe Renal Insufficiency
Brief Title: Liraglutide Treatment to Patients With Severe Renal Insufficiency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bo Feldt-Rasmussen (Other)
Collaborators: Novo Nordisk A/S (Industry); The GCP unit at Copenhagen University Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Bo Feldt-Rasmussen, Professor, DMSc, Head of Department, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-3-2011-032; 2010-021922-36 (EudraCT Number)
Record Dates: First submitted 2011-07-11; First posted 2011-07-14 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Type 2 Diabetes Mellitus; End-stage Renal Disease
Keywords: Liraglutide; Uremia; Dialysis; Type 2 diabetes mellitus; Safety; Efficacy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Kidney Failure, Chronic; Uremia | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- T2D, Dialysis, Liraglutide (Active Comparator): Daily liraglutide treatment Chronic dialysis treatment
  Interventions: Drug: Liraglutide
- T2D, Dialysis, Placebo (Placebo Comparator): Daily placebo Chronic dialysis treatment
  Interventions: Drug: Liraglutide
- T2D, Normal kidney function, Liraglutide (Active Comparator): Daily Liraglutide treatment Normal kidney function
  Interventions: Drug: Liraglutide
- T2D, Normal kidney function, Placebo (Placebo Comparator): Daily placebo treatment Normal kidney function
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Liraglutide — Daily sc. injection, individual dosage
  Other Names: Victoza

SUMMARY:
Incretin-based therapy for the treatment of patients with type 2 diabetes mellitus (T2D) is new and fundamentally different from the classical treatments with oral antidiabetic agents and insulin. The novel and original aspect of this investigator-initiated study is the focus on treatment with an incretin-based agent (the GLP-1 analogue liraglutide) in T2D patients with severely reduced kidney function. At present there is virtually no knowledge of the physiology and clinical implications of the role of incretin hormones and incretin-based therapy in this group of diabetic patients.The aim of the study is to establish an evidence-based rationale for introducing a GLP-1 analogue to the limited armamentarium of antidiabetic drugs for patients with type T2D and severe renal insufficiency. The overall hypothesis is that patients with T2D and severe renal insufficiency will tolerate and benefit from treatment with the GLP-1 analogue liraglutide, hereby improving glycaemic control and reducing risk factors of cardiovascular disease

ELIGIBILITY:
Inclusion criteria - patients with T2D in dialysis

* Male or female; aged 18-85 years
* End-stage renal disease
* Chronic dialysis treatment (minimum 3 months)
* T2D (diagnosed according to WHO criteria)
* Treated with diet/lifestyle intervention, oral antidiabetic drugs (SU, glitazones) and/or insulin
* Documented beta cell function (evaluated by a glucagon test)

Inclusion criteria - patients with T2D and normal kidney function

* Male or female; aged 18-85 years
* Normal kidney function: Plasma creatinine <0.105 mmol/L for men and <0.090 mmol/L for women
* T2D (diagnosed according to WHO criteria)
* Treated with diet/lifestyle intervention, oral antidiabetic drugs (SU, glitazones) and/or insulin
* Documented beta cell function (evaluated by a glucagon test)
* Hemoglobin A1c ≥6.5%

Exclusion Criteria - both groups

* Type 1 diabetes mellitus
* Chronic pancreatitis / previous acute pancreatitis
* Known or suspected hypersensitivity to trial product(s) or related products
* Treatment with oral glucocorticoids, calcineurin inhibitors, dipeptidyl peptidase 4 (DPP4) inhibitors or other drugs, which in the Investigator's opinion could interfere with glucose or lipid metabolism 90 days prior to screening
* Cancer (except basal cell skin cancer or squamous cell skin cancer) or any other clinically significant disorder which in the investigators' opinion could interfere with the results of the trial
* Inflammatory bowel disease
* Cardiac disease defined as: decompensated heart failure (NYHA class III-IV) and/or diagnosis of unstable angina pectoris and/or myocardial infarction within the last 6 months
* Body mass index ≤ 18.5 kg/m2 or ≥ 50.0 kg/m2
* Females of childbearing potential who are pregnant, breast-feeding, intend to become pregnant or are not using adequate contraceptive methods
* Clinical signs of diabetic gastroparesis
* Impaired liver function (transaminases >two times upper reference levels)
* Receipt of any investigational product 90 days prior to this trial
* Known or suspected abuse of alcohol or narcotics
* Screening calcitonin ≥50 ng/l
* Subjects with personal or family history of medullary thyroid carcinoma or a personal history of multiple endocrine neoplasia type 2

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Plasma liraglutide concentration (pmol/L) | 12 weeks
  Plasma liraglutide concentration evaluated over time during continuous intervention

SECONDARY OUTCOMES:
Hypoglycaemia; minor or major | 12 weeks
  Number of hypoglycaemic episodes during intervention. Minor (blood glucose <3.1 mmol/L, no need for assistance). Major (blood glucose <3.1 mmol/L, assistance from third person required)
Glycaemic control | 12 weeka
  Glycaemic control evaluated from 3 daily measurements of blood glucose, from 4 periods of 24-hour tissue glucose measurements (5 days each) and from HbA1c during the intervention period.
Pancreatic beta-cell function | 12 weeks
  Pancreatic beta-cell function evaluated from insulin- and C-peptide-secretion during a standard meal test 3 times during the intervention period.
Cardiovascular risk factors (lipids and blood pressure) | 12 weeks
  Blood pressure will be evaluated at each visit and lipid profile (HDL, LDL, total cholesterol and triglyceride) 3 times during the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Feldt-Rasmussen, Prof, DMSc, Study Director — Department of Nephrology P, Copenhagen University Hospital, Rigshospitalet; Thomas Idorn, MD, Principal Investigator — Department of Nephrology P, Copenhagen University Hospital, Rigshospitalet
Locations (3):
- Denmark (3):
  - Department of Endocrinology PE, Copenhagen University Hospital, Rigshospitalet, Copenhagen Ø, Copenhagen
  - Department of Nephrology P, Copenhagen University Hospital, Rigshospitalet, Copenhagen Ø, Copenhagen
  - Department of Internal Medicine H, Hillerød Hospital, Hillerød

REFERENCES:
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- [Derived] Idorn T, Knop FK, Jorgensen MB, Jensen T, Resuli M, Hansen PM, Christensen KB, Holst JJ, Hornum M, Feldt-Rasmussen B. Safety and Efficacy of Liraglutide in Patients With Type 2 Diabetes and End-Stage Renal Disease: An Investigator-Initiated, Placebo-Controlled, Double-Blind, Parallel-Group, Randomized Trial. Diabetes Care. 2016 Feb;39(2):206-13. doi: 10.2337/dc15-1025. Epub 2015 Aug 17. PMID 26283739
- [Derived] Idorn T, Knop FK, Jorgensen M, Jensen T, Resuli M, Hansen PM, Christensen KB, Holst JJ, Hornum M, Feldt-Rasmussen B. Safety and efficacy of liraglutide in patients with type 2 diabetes and end-stage renal disease: protocol for an investigator-initiated prospective, randomised, placebo-controlled, double-blinded, parallel intervention study. BMJ Open. 2013 Apr 26;3(4):e002764. doi: 10.1136/bmjopen-2013-002764. Print 2013. PMID 23624993